



#### **ASSENT FORM FOR CHILDREN AGES 7 - 11**

Nemours Template December 2024

Your parent has given permission for you to be in a project called a research study. But first, we want to tell you about it so you can decide if you want to be in it. If you don't understand, please ask guestions.

## 1. What is the name of the study?

The Utilization of Ultrasound to Diagnose Pediatric Elbow Fractures: Evaluation of Cost Savings, Radiation Exposure, and Patient Satisfaction

# 2. Who is in charge of the study?

The doctor in charge of the study is Dr. Jason Malone, DO.

### 3. What is the study about?

We would like to find the easiest way to see if you have broken your elbow. There are different types of pictures that the doctor can take to see the inside of your elbow, and they can help tell the doctor if your elbow is hurt. This study is trying to find out if taking one of the types of pictures might hurt less or be easier for you. There are differences between the two types of pictures that this study is using, x-rays and ultrasounds. You might have just one type of picture take of your elbow, or you might have both types taken.

### 4. What will happen to me in the study?

First, the study team will talk to you to make sure you want to be part of this study. The study team will then take a picture of your elbow, with an x-ray or an ultrasound machine. To take an ultrasound picture, the study team will put a wand on the skin of your elbow which only touches your skin a little bit. The study team will also want to talk to you afterwards to find out how you felt about the picture process. If any of the questions that the study team asks you make you uncomfortable or embarrassed, you do not need to answer them. Please talk to the study team if anything about this study makes you uncomfortable. The study team will also want to talk to you in one week, to make sure that your elbow is healing well. You might need to come into the clinic for another exam and x-ray if your elbow is still hurting.

### 5. Do I have to be in the study?

You don't have to do the study if you don't want to. If you are in the study, you can stop being in it at any time. Nobody will be upset with you. No matter what you decide, the doctors and their helpers will take care of you just like they did before. If you have any questions or don't like what is happening, please tell your parent, the doctor or helper.

You have had the study explained to you. You have been given a chance to ask questions. By writing your name below, you are saying that you want to be in the study.



| Name of Child ( <b>Print</b> ) | |
|---|---|
| Signature of Child | Date |
| Name of Person Obtaining Assent ( <b>Print</b> ) | |
| Signature of Person Obtaining Assent | Date |
| The assent information was read to the child by the page of the child read the assent him / herself. | person obtaining assent. |